CLINICAL TRIAL: NCT02193438
Title: Physiologic Effect of Spices Ingestion
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Société des Produits Nestlé (SPN) (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple
Other Study IDs: 10.24.MET
Record Dates: First submitted 2014-07-16; First posted 2014-07-17 (Estimated); Last update posted 2014-07-17 (Estimated); Status verified 2014-07

CONDITIONS: Healthy
Keywords: Heart rate variability; Resting energy expenditure; Facial thermography; Blood pressure; Spices ingestion

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- Spice 1 (Active Comparator): Red chili pepper extract
  Interventions: Other: Placebo
- Spice 2 (Active Comparator): Cinnamon extract
  Interventions: Other: Placebo
- Spice 3 (Active Comparator): Refreshing agent
  Interventions: Other: Placebo
- Placebo (Placebo Comparator): Tomato juice
  Interventions: Other: Spices intake

INTERVENTIONS:
Other: Spices intake — Each subject had to ingest a single dose of each of the spices and placebo. Recording of outcomes was realized throughout the 90 minutes following ingestion.
  Other Names: 3 different spices
  Arms: Placebo
Other: Placebo — Tomato juice intake
  Other Names: Tomato juice
  Arms: Spice 1; Spice 2; Spice 3

SUMMARY:
Human studies have shown that capsaicin, a compound extracted from chilly peppers, can stimulate certain physiologic functions (for example, energy expenditure, thermogenesis, lipid oxidation, heart rate, etc.).

The purpose of this study is to measure the impact of ingesting various spicy molecules on a set of physiologic parameters compared to a placebo. The molecules were selected for their different sensory properties.

The results of this study will allow us to implement an effective method for measuring the impact of ingesting spices on certain body functions (for example, metabolism and autonomic nervous system activity). This study will also allow us to identify the beneficial properties of eating certain spices.

DETAILED DESCRIPTION:
Primary objective and outcome:

The main objective of this study is to establish a methodology to evaluate the acute impact of spice ingestion on metabolism and autonomic nervous system activity.

Primary outcomes:

Impact of the spice on autonomic nervous system activity: Power spectra analysis on heart rate variability (HRV) changes during the 90 post ingestive minutes (measured by ECG).

Impact of the spice on metabolism: Energy expenditure changes during the 90 post ingestive minutes (measured by indirect calorimetry).

As secondary outcomes blood pressure changes and facial temperature changes on specific area (nose, cheeks and forehead) will be evaluated. Substrate oxidation (carbohydrates and fat utilization) and the respiratory quotient (RQ) will be calculated using indirect calorimetry data for energy expenditure measure.

ELIGIBILITY:
Inclusion Criteria:

* Healthy
* BMI: 19-25 kg/m2, ≥ 60 kg body weight
* Moderate spicy food eaters
* Having signed the informed consent.

Exclusion Criteria:

* Any gastrointestinal disorder
* Subject sensitive or not used to eat spicy food
* Smokers
* Subject with beard or mustache
* Abnormal thyroid function
* Intake of medication that could affect body weight and/or energy expenditure
* Weight loss > 5% in the last 3 months
* Under antibiotics or regular treatments (medical or nutritional program) affecting body weight, appetite, energy expenditure, lipid-lowering, hypertension or inflammation or glucose control for the last 3 months or taking hormone replacement therapy
* History of allergy
* Physical activity level > 300 min of moderate or intense exercise per week
* Have a alcohol consumption higher than than 1 drink/day
* Consumption of illicit drugs
* Subject who cannot be expected to comply with the study procedures, including consuming the test products
* Currently participating or having participated in another clinical trial during the last 4 weeks prior to the beginning of this study

Ages: 20 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 19 (Actual)
Dates: Start 2011-05; Primary Completion 2012-08 (Actual); Study Completion 2012-08 (Actual)

PRIMARY OUTCOMES:
Resting energy expenditure | change from baseline to 90 minutes following product intake
  Calculation of the resting energy expenditure from continuous measurement of oxygen consumption and carbon dioxid production (indirect calorimetry).
Heart rate variability | Change from baseline to 90 minutes following product intake
  Power spectral analysis of heart rate variability from continuous measurement of very low, low and high frequency range electrocardiographic signals.

SECONDARY OUTCOMES:
Substrat oxidation | Change from baseline to 90 minutes following product intake
  Carbohydrate oxidation, lipid oxidation, and respiratory quotient from continuous measurements by indirect calorimetryof oxygen consumption and carbon dioxide production.
Blood pressure | every 15 minutes over 90 minutes of recording following product intake
  Standard blood pressure monitoring using an arm cuff
Facial skin temperature modification | Change from baseline to 90 minutes following product intakeover 90 min
  Measurement of the skin temperature of the face using an infrared camera (FLIR A325)

CONTACTS AND LOCATIONS:
Overall Officials: Stéphanie Michlig Gonzalez, PhD, Study Director — Société des Produits Nestlé (SPN); Maurice Beaumont, MD, PhD, Principal Investigator — Société des Produits Nestlé (SPN)
Locations (1):
- NESTEC / Metabolic Unit, Lausanne, Switzerland

REFERENCES:
- [Derived] Tomsen N, Alvarez-Berdugo D, Rofes L, Ortega O, Arreola V, Nascimento W, Martin A, Cabib C, Bolivar-Prados M, Mundet L, Legrand C, Clave P, Michlig S. A randomized clinical trial on the acute therapeutic effect of TRPA1 and TRPM8 agonists in patients with oropharyngeal dysphagia. Neurogastroenterol Motil. 2020 Jun;32(6):e13821. doi: 10.1111/nmo.13821. Epub 2020 Feb 16. PMID 32064725
- [Derived] Michlig S, Merlini JM, Beaumont M, Ledda M, Tavenard A, Mukherjee R, Camacho S, le Coutre J. Effects of TRP channel agonist ingestion on metabolism and autonomic nervous system in a randomized clinical trial of healthy subjects. Sci Rep. 2016 Feb 17;6:20795. doi: 10.1038/srep20795. PMID 26883089